CLINICAL TRIAL: NCT05729984
Title: Comparing Effectiveness of Paula Method Versus Chewing Gum for Postoperative Recovery of Gastrointestinal Function in Patients After Elective Caesarean Section
Brief Title: Paula Method Versus Chewing Gum for Postoperative Recovery After Caesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Joshua Rosenbloom, Attending Physician, Hadassah Medical Organization
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0491-22-HMO
Record Dates: First submitted 2023-01-31; First posted 2023-02-15 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Cesarean Delivery Affecting Fetus; Post Operative Bowel Function
MeSH Terms: interventions — Chewing Gum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paula (Experimental): The patients will perform Paula exercises after cesarean delivery.
  Interventions: Behavioral: Paula exercises
- Gum chewing (Active Comparator): The patients will chew gum after the cesarean delivery.
  Interventions: Behavioral: Gum chewing

INTERVENTIONS:
Behavioral: Paula exercises — The patients will perform Paula exercises after the cesarean delivery
  Arms: Paula
Behavioral: Gum chewing — The patients will be given chewing gum and will be asked to chew it after the cesarean delivery
  Arms: Gum chewing

SUMMARY:
The goal of this clinical trial is to compare the effectiveness of gum chewing vs Paula exercises in patients after cesarean delivery. The main question it aims to answer is: does the Paula method hasten the time to recovery of bowel function compared to gum chewing after cesarean delivery.

Participants will be asked to either chew gum or to do Paula exercises. The time to restoration of bowel function after the surgery will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Women after an elective caesarean delivery
* Age 18+
* Ability to read and write in Hebrew

Exclusion Criteria:

* Diagnosis of chronic gastrointestinal diseases
* Inability to chew gum
* Use of laxatives.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2023-05-24 (Actual); Study Completion 2023-05-24 (Actual)

PRIMARY OUTCOMES:
Time to first flatus or bowel movements | Up to one week from delivery
  The patients will note the time of the first passing gas and the first bowel movement after the cesarean delivery.

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No